CLINICAL TRIAL: NCT00966511
Title: Vibration Response Imaging (VRI) in Patients Who Are Potential Candidates for Surgical Resection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat / VP Clinical Affairs, Deep Breeze
Other Study IDs: DB041
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; lung resection; lobectomy; pneumonectomy; lung function; perfusion
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung resection candidates: Study participants will be patients who are candidates for lung resection (lobectomy or greater)
  Interventions: Procedure: Lung resection surgery

INTERVENTIONS:
Procedure: Lung resection surgery — The study is designed in a way that will not alter the surgeon's decision based on routine assessment of candidates for resection (lobectomy or greater). Namely, the VRI data will be gathered prospectively; however, the analyses using VRI data will be performed retrospectively.

SUMMARY:
The primary purpose of the study is to investigate the use of VRI to guide the selection of patients for lung surgery. Perfusion scintigraphy is the current method to assess the fractional contribution of lung function of the remaining lung.

The hypothesis is that VRI can determine quantitative postoperative lung function equally accurately as a quantitative perfusion scan.

DETAILED DESCRIPTION:
Primarily, VRI will be compared to perfusion (Q) scan by predicted post-operative (ppo) FEV1 and DLCO as predicted by VRI versus as predicted by Q scan. Secondary, the ppo as predicted by each test will be compared with the actual FEV1 and DLCO at 3 months post-operative; If these two methods provide similar results, VRI will be deemed an acceptable alternative to Q scan for determining patient selection for lung resection. Finally, the patient outcomes (30 day mortality and pulmonary complications) for those patients falling within guideline parameters using the VRI measurement will be analyzed to see if using VRI in clinical practice would indeed allow prediction of satisfactory results (similar to literature benchmarks).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to read, understand, and provide written Informed Consent;
2. Age range of 18-90 years;
3. Potential candidate for at least lobectomy due to lung cancer or other intrathoracic malignancy (either suspected or proven by biopsy). Both open and minimally invasive (thoracoscopic) resections are acceptable.
4. BMI > 19.

Exclusion Criteria:

1. Body habitus or skin condition that might prevent the placement of the sound sensors on the back (e.g. severe scoliosis, kyphosis, chest wall deformation, skin lesion on the back or compression fracture);
2. There should be no active pulmonary infection (e.g. pneumonia) at the time of the recordings;
3. Hirsutism unless patient is willing to have back shaved;
4. Potentially contagious skin lesion on the back;
5. Giant bulla (more than 1/3 of the hemithorax or >10cm)
6. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be patients who are candidates for lung resection (lobectomy or greater)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of ppo FEV1 and ppo DLCO as predicted by VRI with the values as predicted by Q scan | Prior to surgery

SECONDARY OUTCOMES:
Comparison of ppo as predicted by each test with the actual FEV1 and DLCO at 3 months post-operative | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank C Detterbeck, MD, Principal Investigator — Yale University Medical School
Locations (6):
- United States (6):
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston University, Boston, Massachusetts
  - Mt. Sinai School of Medicine, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Dellinger RP, Parrillo JE, Kushnir A, Rossi M, Kushnir I. Dynamic visualization of lung sounds with a vibration response device: a case series. Respiration. 2008;75(1):60-72. doi: 10.1159/000103558. Epub 2007 Jun 4. PMID 17551264
- [Background] Kramer MR, Raviv Y, Hardoff R, Shteinmatz A, Amital A, Shitrit D. Regional breath sound distribution analysis in single-lung transplant recipients. J Heart Lung Transplant. 2007 Nov;26(11):1149-54. doi: 10.1016/j.healun.2007.07.039. PMID 18022081
- [Background] Yigla M, Gat M, Meyer JJ, Friedman PJ, Maher TM, Madison JM. Vibration response imaging technology in healthy subjects. AJR Am J Roentgenol. 2008 Sep;191(3):845-52. doi: 10.2214/AJR.07.3151. PMID 18716118
- [Background] Guntupalli KK, Reddy RM, Loutfi RH, Alapat PM, Bandi VD, Hanania NA. Evaluation of obstructive lung disease with vibration response imaging. J Asthma. 2008 Dec;45(10):923-30. doi: 10.1080/02770900802395496. PMID 19085584
- [Background] Becker HD, Slawik M, Miyazawa T, Gat M. Vibration response imaging as a new tool for interventional-bronchoscopy outcome assessment: a prospective pilot study. Respiration. 2009;77(2):179-94. doi: 10.1159/000182972. Epub 2008 Dec 9. PMID 19065052
- [Background] Colice GL, Shafazand S, Griffin JP, Keenan R, Bolliger CT; American College of Chest Physicians. Physiologic evaluation of the patient with lung cancer being considered for resectional surgery: ACCP evidenced-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):161S-77S. doi: 10.1378/chest.07-1359. PMID 17873167